CLINICAL TRIAL: NCT06939374
Title: Clinical Investigation of the Efficacy and Safety of Intracoronary Cryotherapy Using the CryoTherapy System (CTS) for High-risk Plaque in Patients With Stable Angina or Acute Coronary Syndrome.
Brief Title: Intracoronary Cryotherapy Effect on Stabilization of Vulnerable Plaque in Patients With Stable Angina or ACS - A Traditional Feasibility Study
Acronym: ICECAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cryotherapeutics SA (Industry)
Collaborators: CoreAalst BV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-CP-P01_0104
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Coronary Arterial Disease (CAD); Plaque; Vulnerable Plaque; Cryotherapy; Cryotherapy Effect; Coronary Balloon; Atherosclerosis Coronary Artery With Angina Pectoris
Keywords: Medical device; traditional feasibility; Single Group; Device Feasibility; Multi-Center; Prospective; Interventional
MeSH Terms: conditions — Plaque, Amyloid

STUDY DESIGN:
Intervention Model Description: Prospective, Multi-Center, Interventional, Device Feasibility
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Subjects with coronary HRP lesions treated with intracoronary cryotherapy using the CTS device
  Interventions: Device: Intracoronary Cryotherapy

INTERVENTIONS:
Device: Intracoronary Cryotherapy — Intracoronary cryotherapy for stabilization of High-risk coronary plaque

SUMMARY:
ICECAP is a multi-centre, prospective, single-arm, interventional, traditional feasibility clinical investigation to evaluate the efficacy and safety of intra-coronary cryotherapy on vulnerable or high-risk plaque (HRP), using the CryoTherapy System (CTS). The study aims to enroll 25 patients with symptomatic coronary artery disease, successfully treated for their culprit lesion and with presence of at least one HRP lesion in another vessel. Eligible patients will undergo cryotherapy during a planned procedure. Near-infrared spectrometry (NIRS and Optical Coherence Tomography imaging will be used during baseline procedure, and during a 9 months follow visit. The primary endpoint is reduction of plaque burden measured as 30% reduction in maxLCBI4mm as measured by NIRS at 9 months post procedure.

DETAILED DESCRIPTION:
ICECAP is a multi-centre, prospective, single-arm, interventional, traditional feasibility clinical investigation to evaluate the efficacy and safety of intra-coronary cryotherapy on vulnerable or high-risk plaque (HRP), using the CryoTherapy System (CTS). The study aims to enroll 25 patients with stable angina or Acute Coronary Syndrome (ACS). Patients who have undergone successful treatment of their culprit lesion, and in whom presence of at least one non-flow-limiting HRP lesion in another vessel is identified (confirmed by Coronary Computed Tomography Angiography - CCTA), are eligible for the study. Eligible patients will undergo cryotherapy using the CTS during a planned procedure within maximum 8 weeks after eligibility has been confirmed. Near-infrared spectrometry (NIRS) and Optical Coherence Tomography (OCT) imaging will be used during baseline procedure, and during a 9 months angiographic follow visit. Clinical follow-up visits will be done at 1, 3, 6, 9 and 12 months post-procedure. The primary endpoint is reduction of plaque burden, defined as 30% reduction in maxLCBI4mm measured by NIRS at 9 months post procedure. Secondary efficacy endpoints include: changes in fibrous cap thickness assessed by OCT at 9 months post-procedure, changes in Plaque volume and plaque composition at 9 months post-procedure. Safety endpoints include procedural success rates, any cryotherapy related complication or any Major Adverse Cardiac Event (MACE) at 3 and 12 months post procedure. The enrolment period is expected to last 9 months, and all subjects will be followed for 12 months after the CTS procedure.

ELIGIBILITY:
Inclusion Criteria:

* 1) Subject is at least 18 years old. 2) Subject has acute cardiac pain/angina consistent with stable angina or acute coronary syndrome eligible for coronary angiography meeting one of the following criteria:

  1. Non-ST-segment elevation myocardial infarction (NSTEMI) with rise/fall of cardiac enzymes (troponin I or T) with at least one value above the 99th percentile of the upper reference limit requiring PCI within 72 hours from diagnosis
  2. Unstable angina
  3. ST-segment elevation myocardial infarction (STEMI) 3) Successful PCI (defined as diameter stenosis less than 30% and TIMI 3 flow on final angiography without procedural complication) of the culprit lesion.

NOTE: subjects with unstable angina, for whom the culprit lesion as assessed by investigator does not require PCI currently or within the next 6 months (subject treated with optimal medical treatment) can be enrolled in the study.

4) Subject has at least one high-risk plaque meeting the criteria below:

1. Located in a non-culprit vessel,
2. High-risk plaque lesion on CCTA and at least one of the following features:

   1. Presence of low-attenuation plaque (HU<50) and/or
   2. Positive remodelling (remodelling index >1.1) and/or
   3. Napkin ring sign and/or
   4. Plaque burden ≥70%
3. Lesion length ≤ 20 mm.
4. Diameter stenosis on invasive angiography between 30% and 70% on coronary angiogram or negative physiology assessment (FFR>0.80 or NHPR>0.89).
5. Reference vessel diameter (RVD) < 3.75 mm and > 2.50 mm in diameter
6. Investigator considers that lesions are accessible.
7. If more than two suitable lesions available, investigator will select the most appropriate lesion for cryotherapy treatment.

   5) maxLCBI4mm in the lesion > 324.7 6) Subject is able to provide consent and has signed and dated the informed consent form.

   Exclusion Criteria:
   * 1) Subject is hemodynamically unstable (cardiogenic shock, hypotension needing inotropes, hypoxia needing intubation, refractory ventricular arrhythmias, and IABP).

     2) Subject has ongoing ST-segment elevation myocardial infarction. 3) Subject had a procedural complication during the ACS PCI procedure. 4) Subject has history of Coronary Artery Bypass Graft (CABG) or planned CABG within 12 months after the index procedure.

     5) Subject has known reduced Left Ventricular Ejection Fraction < 30%. 6) Subject has known severe valvular heart disease. 7) Subject has known severe renal insufficiency (eGFR <30 ml/min/1.72 m2). 8) Subject has any life-threatening conditions or medical comorbidity resulting in life expectancy < 12 months.

     9) Subject is currently participating in another clinical investigation that has not yet reached its primary endpoint.

     10) Subject has severe peripheral vascular disease impeding femoral artery access.

     11) Subject is pregnant or lactating, or NOT surgically sterile (tubal ligation or hysterectomy) or NOT postmenopausal for at least 6 months or is a female with childbearing potential without effective contraception (pill, patch, ring, diaphragm, implant and intrauterine device).

   Angiographic exclusion criteria:
   1. Visible distal embolization/no-reflow following culprit lesions PCI.
   2. Left main coronary artery disease (visual diameter stenosis > 50%).
   3. Stent thrombosis/restenosis as a culprit lesion.
   4. CTS lesion involving a bifurcation (defined as lesions involving side branches >2.0 mm).
   5. Angiographic or CCTA evidence of severe calcification and/or marked tortuosity of the index vessel and/or lesion.
   6. Thrombotic lesions.
   7. Ostial lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in MaxLCBI4mm | At 9 months post-CTS procedure compared to baseline.
  Reduction of at least 30% in maxLCBI4mm in the lesion measured by NIRS

SECONDARY OUTCOMES:
Change in Fibrous Cap Thickness | At 9 months post-CTS procedure compared to baseline
  Change in OCT-derived fibrous cap thickness
Change in Minimal Lumen Area (MLA) | At 9 months post-CTS procedure compared to baseline.
  Change in minimum lumen area (MLA) by OCT
Prevalence of Thin Cap Fibrous Atheroma | At 9 months post-CTS procedure compared to baseline.
  Prevalence of thin cap fibroatheroma (minimum fibrous cap thickness < 65 µm with lipid arc > 90°) by OCT.
Prevalence of lipid Arc >90° | At 9 months post-CTS procedure compared to baseline.
  Prevalence of lipid arc greater than 90° by OCT.
Prevalence of lipid Arc >180° | At 9 months post-CTS procedure compared to baseline.
  Prevalence of lipid arc greater than 180° by OCT.
Prevalence of lipid Arc >270° | At 9 months post-CTS procedure compared to baseline.
  Prevalence of lipid arc greater than 270° by OCT.
Total angle of macrophage | At 9 months post-CTS procedure compared to baseline.
  Total angle of macrophage within the treated segment by OCT.
Maximum angle of macrophage | At 9 months post-CTS procedure compared to baseline.
  Maximum angle of macrophage within the treated segment by OCT.
Total angle of lipidic plaque | At 9 months post-CTS procedure compared to baseline.
  Total angle of lipidic plaque within the treated segment by OCT.
Maximum angle of lipidic plaque | At 9 months post-CTS procedure compared to baseline.
  Maximum angle of lipidic plaque within the treated segment by OCT.
Total angle of calcification | At 9 months post-CTS procedure compared to baseline.
  Total angle of calcification within the treated segment by OCT.
Maximum angle of calcification | At 9 months post-CTS procedure compared to baseline.
  Maximum angle of calcification within the treated segment by OCT.
Total Plaque volume | At 12 months post-CTS procedure compared to baseline.
  Total Plaque volume within the treated lesion segment assessed by CCTA
Calcified Plaque volume | At 12 months post-CTS procedure compared to baseline.
  Calcified Plaque volume within the treated lesion segment assessed by CCTA
Area stenosis | At 12 months post-CTS procedure compared to baseline.
  Area stenosis within the treated lesion segment assessed by CCTA

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Collet, MD, Study Chair — AZORG Hospital, Aalst, belgium

IPD SHARING:
Plan to Share IPD: No